CLINICAL TRIAL: NCT04447352
Title: Preventive HIPEC in Combination With Perioperative FLOT Versus FLOT Alone for Resectable Diffuse Type Gastric and Gastroesophageal Junction Type II/III Adenocarcinoma - The Phase III "PREVENT" Trial of the AIO /CAOGI /ACO
Brief Title: HIPEC + FLOT vs. FLOT Alone in Patients With Gastric Cancer and GEJ (PREVENT)
Acronym: PREVENT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Krankenhaus Nordwest (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIPEC/FLOT9; AIO-STO-0319/ass (Other: AIO number)
Record Dates: First submitted 2020-06-17; First posted 2020-06-25 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - FLOT (Active Comparator): Patients randomized to treatment Arm A already received 3-6 cycles of FLOT in 2-week treatment cycles prior to undergoing surgery. Following surgery, patients will receive four further 2-week cycles FLOT. FLOT can be deescalated to FLO, FLT or FL in case of chemorelated toxicity at any time and at the discretion of investigator.
  FLOT = Docetaxel 50 mg/m², Oxaliplatin 85 mg/m², Leucovorin 200 mg/m², 5-FU 2600 mg/m².
  Interventions: Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Docetaxel
- Arm B - FLOT/HIPEC (Experimental): Patients randomized to treatment Arm B already received 3-6 cycles of FLOT in 2-week treatment cycles prior to undergoing surgery including Intraoperative Hyperthermic IntraPEritoneal Chemoperfusion (HIPEC) during gastric-/ esophagogastric resection using Cisplatin 75mg/m². Following surgery, patients will receive four further 2-week cycles FLOT. FLOT can be deescalated to FLO, FLT or FL in case of chemorelated toxicity at any time and at the discretion of investigator.
  FLOT = Docetaxel 50 mg/m², Oxaliplatin 85 mg/m², Leucovorin 200 mg/m², 5-FU 2600 mg/m².
  Interventions: Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Docetaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: 5-Fluorouracil — Day 1 q2w: 2600 mg/m² IV over 24 hours
  Other Names: 5-FU
Drug: Leucovorin — Day 1 q2w: 200 mg/m² IV over 30 minutes
  Other Names: Calciumfolinat
Drug: Oxaliplatin — Day 1 q2w: 85 mg/m² IV over 2 hours
Drug: Docetaxel — Day 1 q2w: 50 mg/m² IV over 1 hour
Drug: Cisplatin — intraoperative: 75mg/m² intraabdominal solution over 1 hour and 30 minutes
  Arms: Arm B - FLOT/HIPEC

SUMMARY:
This is a multicenter, randomized, controlled, open-label study evaluating efficacy and safety of perioperative FLOT chemotherapy plus intraoperative HIPEC versus FLOT chemotherapy alone in patients with resectable localized and locally advanced diffuse and mixed type adenocarcinoma of the stomach and Type II/III GEJ.

DETAILED DESCRIPTION:
This is a multicenter, randomized, controlled, open-label study including patients with localized and locally advanced diffuse and mixed type adenocarcinoma of the stomach and Type II/III GEJ scheduled to receive perioperative chemotherapy combined with intraoperative HIPEC procedure.

The scope of the trial is to evaluate the efficacy as well as the safety and tolerability of the combination of perioperative chemotherapy combined with an intraoperative HIPEC for resectable diffuse and mixed type gastric and GEJ (types II/III) adenocarcinoma. Intraoperative hyperthermic chemoperfusion is summarized under the abbreviation HIPEC in the following.

Patients with localized and locally advanced diffuse or mixed type adenocarcinoma of the stomach and Type II/III GEJ (i.e. ≥cT3 any N or any T N-positive) with exclusion of distant metastases and after receiving neoadjuvant FLOT- therapy will be included in this trial after a central review.

All enrolled patients will have received 3-6 pre-operative cycles (de-escalation or dose modification allowed) of biweekly FLOT (Docetaxel 50 mg/m² in 250 ml NaCl 0.9%, iv over 1 h; Oxaliplatin 85 mg/m² in 500 ml G5%, iv over 2h; Leucovorin 200 mg/m² in 250 ml NaCl 0.9%, iv over 30 min; 5-FU 2600 mg/m², iv over 24 h, q2wk) in the preoperative treatment phase.

After completion of neoadjuvant FLOT- therapy followed by pre-operative tumor assessment, (also including diagnostic laparoscopy prior to start of FLOT), patients without disease progression (expected to be approximately 90% of the patients) will be included into the trial, stratified by initial clinical stage (N- vs. N+), histological type of tumor (Lauren classification diffuse vs. mixed) and study site.

Patients will be randomized 1:1 to receive either postoperative FLOT (Arm A) or postoperative FLOT + intraoperative HIPEC (Arm B).

Arm A (FLOT) Surgery in Arm A is planned to occur 4 to 6 weeks after d1 of last FLOT. Surgery is carried out in kind of gastrectomy, transhiatal extended gastrectomy. Following surgery, patients will receive four further 2-week treatment cycles FLOT in the post-operative treatment phase. Post-operative treatment should start 6 to 8 weeks, but at maximum 12 weeks after surgery.

Arm B (FLOT/ HIPEC) Surgery in Arm B is planned to occur 4 to 6 weeks after d1 of last FLOT. Surgery is carried out in kind of gastrectomy, transhiatal extended gastrectomy. Surgery will be combined with an intraoperative Hyperthermic IntraPEritoneal Chemoperfusion (HIPEC) including cisplatin solution administered at a temperature of 42°C for 90 minutes. Following surgery, patients will receive four further 2-week treatment cycles FLOT in the post-operative treatment phase. Post-operative treatment should start 6 to 8 weeks, but at maximum 12 weeks after surgery.

In both of the arms, tumor assessments (CT or MRI) are performed before randomization prior to surgery, and then every 3 months (radiological tumor assessment) thereafter until progression/relapse, death or end of follow-up. A change from CT into MRI in the follow up period is possible at any time.

During treatment, clinical visits (blood cell counts, detection of toxicity) occur prior to every treatment dose. Safety of FLOT/ HIPEC will be monitored continuously by careful monitoring of all adverse events (AEs) and serious adverse events (SAEs) reported.

The phase III design starts with a safety run-in phase. After 20 patients had curatively intended resection in Arm B, an interim safety analysis is performed that shows feasibility, safety, and tolerability of Arm B planned at the time 8 weeks after the 20th patient in Arm B had curatively intended resection. It is not planned to discontinue recruitment for the interim safety analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed, medically operable, resectable diffuse or mixed type (according to Lauren's classification) adenocarcinoma of the gastroesophageal junction (AEG II-III) or the stomach (uT3, uT4a, any N category, M0), or any T N+ M0 patient
2. Patient has received 3 to 6 cycles of neoadjuvant FLOT (de-escalation or dose modification allowed)
3. No preceding cytotoxic or targeted therapy other than neoadjuvant FLOT (including de-escalated or dose reduced schema) therapy
4. No prior partial or complete tumor resection
5. Female and male patient ≥ 18 and ≤ 75 years. Female patient with childbearing potential needs to have a negative pregnancy test within 7 days prior to study start. Males and females of reproductive potential must agree to practice highly effective contraceptive measures* during the study. Male patients must also agree to refrain from father a child during treatment and additionally to use a condom during treatment period. Their female partner of childbearing potential must also agree to use an adequate contraceptive measure.

   *highly effective (i.e. failure rate of <1% per year when used consistently and correctly) methods: intravaginal and transdermal combined (estrogen and progestogen containing) hormonal contraception; injectable and implantable progestogen-only hormonal contraception; intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner; sexual abstinence (complete abstinence is defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments).
6. ECOG ≤ 1
7. Exclusion of distant metastases by CT or MRI of abdomen, pelvis, and thorax, bone scan or MRI (if bone metastases are suspected due to clinical signs). Exclusion of the infiltration of any adjacent organs or structures by CT or MRI
8. Laparoscopic exclusion of peritoneal carcinomatosis at initial staging, before start of FLOT chemotherapy
9. Hematological, hepatic and renal function parameters adequate to allow surgical procedure and HIPEC at investigator´s discretion
10. Patient able and willing to provide written informed consent and to comply with the study protocol and with the planned surgical procedures

Exclusion Criteria:

1. Patient without neoadjuvant therapy or those who received a neoadjuvant therapy other than FLOT
2. Known hypersensitivity against 5-FU, leucovorin, oxaliplatin, or docetaxel
3. Other known contraindications against, 5-FU, leucovorin, oxaliplatin, or docetaxel
4. Clinically significant active coronary heart disease, cardiomyopathy or congestive heart failure, NYHA III-IV
5. Clinically significant valvular defect
6. Past or current history of other malignancies not curatively treated and without evidence of disease for more than 3 years, except for curatively treated basal cell carcinoma of the skin and in situ carcinoma of the cervix
7. Criteria of primary unresectability, e.g.:

   * Radiologically documented evidence of major blood vessel invasion or invasion of adjacent organs (T4b).
   * Patients with involved retroperitoneal (e.g. para-aortal, paracaval or interaortocaval lymph nodes) or mesenterial lymph nodes (distant metastases!)
8. Other severe internal disease or acute infection
9. Patient has undergone major surgery within 28 days prior to enrollment
10. Cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) and a history of hepatic encephalopathy or ascites.
11. On-treatment participation in another interventional clinical study in the period 30 days prior to inclusion and during the study
12. Patient pregnant or breast feeding, or planning to become pregnant
13. Patient in a closed institution according to an authority or court decision (AMG § 40, Abs. 1 No. 4)
14. Any other concurrent antineoplastic treatment including irradiation
15. Known intraabdominal adhesion situs
16. Pre-existing peritoneal seeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of progression-/disease-free survival (PFS/DFS) between arms | from randomization up to 5 years
  To compare PFS/DFS in patients with localized and advanced diffuse or mixed type adenocarcinoma of the stomach and Type II/III GEJ (i.e. ≥cT3 any N or any T N-positive) with exclusion of distant metastases and after receiving neoadjuvant FLOT- therapy will be included in this trial after a central review, receiving 3-6 cycles perioperative FLOT versus FLOT alone in the intent to treat population (ITT) and where PFS/DFS is defined as the time from randomization to disease progression or relapse after surgery or death from any cause.

SECONDARY OUTCOMES:
Comparison of Overall survival (OS) in both arms | from randomization up to 5 years
  Overall survival (OS) where OS is defined as the time from randomization to death from any cause.
Comparison of Overall survival rates at 3 and 5 years in both arms | 3 and 5 years after randomization
  OS rates at 3 & 5 years defined as the percentage patients known to be alive after 3 and 5 years referring to the total number of patients randomized into the respective treatment arm
Comparison of peritoneal relapse rate at 2 and 3 years in both arms | 2 and 3 years after surgery
  Peritoneal relapse rate defined as the percentage of patients with peritoneal relapse referring to the total number of patients randomized into the respective treatment arm
PFS/DFS rates at 2, 3 & 5 years | 2, 3 & 5 years after randomization
  PFS/DFS rates at 2, 3 & 5 years defined as the percentage of patients without disease progression or relapse after surgery or death from any cause after 2, 3 and 5 years referring to the total number of patients randomized into the respective treatment arm
Rate of surgical serious adverse events (SAEs) | After randomization of the patient until 30 days after last study-specific treatment
  Rate of surgical serious adverse events, according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE Version 5.0) grade ≥ 3 adverse events and grade ≥ 3 laboratory toxicities.
OS and PFS/DFS (medians and rates) according to subgroup (diffuse vs. mixed and gastric vs. GEJ type II/III) | from randomization up to 5 years
  PFS/DFS is defined as the time from randomization to disease progression or relapse after surgery or death from any cause and OS is defined as the time from randomization to death from any cause. OS and PFS/DFS rates are defined as the percentage of patients known to be alive or without disease progression or relapse after surgery or death from any cause, respectively, at specific timepoints and referring to the total number of patients in defined subgroups (diffuse vs. mixed and gastric vs. GEJ type II/III).
Patient reported outcomes: Quality of life EORTC QLQ C30 questionnaire | From date of screening until the date of first documented progression or last visit before date of death from any cause, whichever came first, assessed 8 weeks +/- 7 days until EOT, afterwards every 3 months up to 2 years after last patient in
  The QoL analyses will include QoL mean values, QoL response and time to symptom deterioration (TTSD) defined as the time interval between randomization and the first decrease by ≥ 10-points. All randomly assigned patients with a baseline and at least one post-baseline assessment will be included in TTSD analyses. Patients without observed deterioration will be censored at the time of their last QoL assessment. Questionnaires given to the patients (validated quality of life questionnaires EORTC QLQ C30).
  EORTC QLQ C30 contains 30 questions:
  28 questions regarding body fitness, daily routines, restrictions at work and hobby, appetite, fatigue, cough, breathlessness, pain, tiredness, and body conditions from (1) to (4); 1 (not a bit), 2 (little), 3 (moderate), 4 (much).
  2 questions regarding state of health and Quality of life with a horizontal rating from 1 to 7; 1 (very bad), 7 (excellent).
Patient reported outcomes: Quality of life EORTC QLQ STO22 questionnaire | From date of screening until the date of first documented progression or last visit before date of death from any cause, whichever came first, assessed 8 weeks +/- 7 days until EOT, afterwards every 3 months up to 2 years after last patient in
  The QoL analyses will include QoL mean values, QoL response and time to symptom deterioration (TTSD) defined as the time interval between randomization and the first decrease by ≥ 10-points. All randomly assigned patients with a baseline and at least one post-baseline assessment will be included in TTSD analyses. Patients without observed deterioration will be censored at the time of their last QoL assessment. Questionnaires given to the patients (validated quality of life questionnaires EORTC QLQ STO22).
  The EORTC QLQ-STO 22 module contains 22 items in a similar layout and response format to the EORTC QLQ-C30. The hypothesised scale structure of the module consists of five scales (dysphagia, eating restrictions, pain, reflux and anxiety) and three single items (dry mouth, body image and hair loss).
Patient reported outcomes: VAS pain assessment form | From date of screening until the date of first documented progression or last visit before date of death from any cause, whichever came first, assessed 8 weeks +/- 7 days until EOT, afterwards every 3 months up to 2 years after last patient in
  The patient´s assessment of their current level of pain on a 100-mm horizontal VAS. The left-hand extreme of the line should be described as "no pain" and the right-hand as "unbearable pain".
Rate of post-operative morbidity/mortality at day 30 after surgery acc. to Clavien-Dindo classification | at day 30 after surgery
  Rate of post-operative morbidity/mortality will be assessed at day 30 after surgery acc. to Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten O Götze, MD, Principal Investigator — Lead Coordinating Investigator
Locations (15):
- Germany (15):
  - Uniklinik RWTH Aachen, AöR, Medizinische Klinik III, Studienzentrum Viszeralmedizin, Aachen
  - Universitätsklinikum, Klinik und Poliklinik für Viszeral-, Thorax- und Gefäßchirurgie, Dresden
  - Institute of Clinical Cancer Research (IKF), UCT - University Cancer Center, Frankfurt, Germany, Frankfurt
  - Universitätsklinikum Halle (Saale), Universitätsklinik und Poliklinik für Viszerale, Gefäß- und Endokrine Chirurgie, Halle
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Viszeral-, Transplantations-, Thorax- und Gefäßchirurgie, Leipzig
  - Klinikum Ludwigsburg, Klinik für Innere Medizin, Gastroenterologie, Hämato-Onkologie, Pneumologie, Diabetologie und Infektiologie, Ludwigsburg
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Klinik für Chirurgie, Lübeck
  - Universitätsklinikum Magdeburg, Magdeburg
  - Klinikum rechts der Isar der TU München, Klinik und Poliklinik für Innere Medizin III, München
  - Universitätsklinikum Münster, Klinik für Allgemein-, Viszeral- und Transplantationschirurgie, Münster
  - Krankenhaus Barmherzige Brüder Regensburg, Klinik für Onkologie und Hämatologie, Regensburg
  - Klinikum Südstadt Rostock, Klinik für Innere Medizin III, Rostock
  - Universitätsklinikum Tübingen, Universitätsklinik für Allgemeine, Viszeral- und Transplantationschirurgie Chirurgische Studienzentrale, Tübingen
  - Marien-Hospital Witten, Witten
  - Universitätsklinikum Würzburg, Chirurgische Klinik I, Chirurgisches Studienzentrum, Würzburg

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

REFERENCES:
- [Derived] Gotze TO, Piso P, Lorenzen S, Bankstahl US, Pauligk C, Elshafei M, Amato G, Reim D, Bechstein WO, Konigsrainer A, Monig SP, Rau B, Schwarzbach M, Al-Batran SE. Preventive HIPEC in combination with perioperative FLOT versus FLOT alone for resectable diffuse type gastric and gastroesophageal junction type II/III adenocarcinoma - the phase III "PREVENT"- (FLOT9) trial of the AIO /CAOGI /ACO. BMC Cancer. 2021 Oct 29;21(1):1158. doi: 10.1186/s12885-021-08872-8. PMID 34715810